CLINICAL TRIAL: NCT02621021
Title: A Phase II Trial for Metastatic Melanoma Using Adoptive Cell Therapy With Tumor-Infiltrating Lymphocytes Plus IL-2 Either Alone or Following the Administration of Pembrolizumab
Brief Title: A Phase 2 Trial for Metastatic Melanoma Using Adoptive Cell Therapy With Tumor Infiltrating Lymphocytes Plus IL-2 Either Alone or Following the Administration of Pembrolizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160027; 16-C-0027
Record Dates: First submitted 2015-12-02; First posted 2015-12-03 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-07-08

CONDITIONS: Melanoma
Keywords: Melanoma; Skin Cancer; Immunotherapy; Cell Therapy
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — pembrolizumab; aldesleukin; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1/ACT TIL (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +young TIL + highdose aldesleukin (IL-2)
  Interventions: Biological: young TIL; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide
- 2/ACT TIL + Pembro (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +young TIL + highdose aldesleukin (IL-2) + pembrolizumab
  Interventions: Biological: young TIL; Drug: Pembrolizumab; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide
- 3/ACT TIL (Pembro contraindicated) (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine + young TIL + highdose aldesleukin (IL-2)
  Interventions: Biological: young TIL; Drug: Aldesleukin; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: young TIL — Day 0: Cells will be administered intravenously (IV) on the Patient Care Unit over 20-30 minutes.
Drug: Pembrolizumab — (Cohort 1, Arm 2 ,Cohort 2 and Cohort 3, Arm 2) On day -2, and days 21 (+/- 2 days), 42 (+/- 2 days), and 63 (+/- 2 days) following cell infusion: Pembrolizumab 2mg/kg IV over approximately 30 minutes.
  Arms: 2/ACT TIL + Pembro
Drug: Aldesleukin — Aldesleukin 720,000 IU/kg IV (based on total body weight) over 15 minutes approximately every 8 hours (+/- 1 hour) beginning within 24 hours of cell infusion and continuing for up to 4 days (maximum 12 doses).
Drug: Fludarabine — Days -7 to -3, Fludarabine 25 mg/m2/day IVPB daily over 15-30 minutes for 5 days.
Drug: Cyclophosphamide — Days -7 and -6: Cyclophosphamide 60 mg/kg/day X 2 days IV in 250 ml D5W with mesna 15 mg/kg/day over 1 hour X 2 days.

SUMMARY:
Background:

Cell therapy is an experimental cancer therapy. It takes young tumor infiltrating lymphocytes (Young TIL) cells from a person s tumors and grows them in a lab. Then they are returned to the person. Researchers think adding the drug pembrolizumab might make the therapy more effective.

Objective:

To test if adding pembrolizumab to cell therapy is safe and effective to shrink melanoma tumors.

Eligibility:

People ages 18-72 years with metastatic melanoma OF THE SKIN

Design:

Participants will be screened with:

Physical exam

CT, MRI, or PET scans

X-rays

Heart and lung function tests if indicated

Blood and urine tests

Before treatment, participants will have:

A piece of tumor taken from a biopsy or during surgery in order to grow TIL cells

Leukapheresis: Blood flows through a needle in one arm and into a machine that removes white blood cells.

The rest of the blood returns through a needle in the other arm.

An IV catheter placed in the chest for getting TIL cells, aldesleukin, and pembrolizumab (if assigned)

Participants will stay in the hospital for treatment. This includes:

Daily chemotherapy for 1 week

For some participants, pembrolizumab infusion 1 day after chemotherapy

TIL cell infusion 2-4 days after chemotherapy, then aldesleukin infusion every 8 hours for up to 12 doses

Filgrastim injections to help restore your blood counts

Recovery for 1-3 weeks

After treatment, participants will:

Take an antibiotic and an antiviral for at least 6 months, as applicable

If assigned, have pembrolizumab treatment every 3 weeks for 3 more doses. They may have another round.

Have 2-day follow-up visits every 1-3 months for 1 year and then every 6 months

DETAILED DESCRIPTION:
Background:

- Adoptive cell therapy (ACT) using autologous tumor infiltrating lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting

preparative regimen consisting of cyclophosphamide and fludarabine.

- Pembrolizumab, a monoclonal antibody that binds to PD-1 and blocks the PD-1/PD-L1 axis, facilitates the activity of anti-tumor lymphocytes in the tumor micro environment. Pembrolizumab administration can result in objective tumor responses in patients with

metastatic melanoma and is approved for use by the FDA for the treatment of these patients.

* Administered TIL express low levels of PD-1, though PD-1 can be re-expressed on TIL in vivo following TIL administration.
* In pre-clinical models, the administration of an anti-PD1 antibody enhances the anti-tumor activity of transferred T-cells.

Objectives:

Primary Objectives:

Determine the objective response rate with the addition of

pembrolizumab to the standard non-myeloablative conditioning regimen, TIL, and

high-dose IL-2 in patients with metastatic melanoma who have received prior anti-

PD-1/PD-L1 therapy (Cohorts 1 and 3).

Eligibility:

* Age greater than or equal to 18 and less than or equal to 72 years
* Evaluable metastatic melanoma
* Metastatic melanoma lesion suitable for surgical resection for the preparation of TIL
* No allergies or hypersensitivity to high-dose aldesleukin administration
* No concurrent major medical illnesses or any form of immunodeficiency

Design:

* Patients with metastatic melanoma will have lesions resected for TIL
* Patients will be assigned one of 3 cohorts: (1) patients who are refractory to prior

anti-PD-1/PD-L1 therapy (randomized); (2) patients who have not received prior anti-

PD-1/PD-L1 therapy; and (3) patients who are refractory to anti PD-1/PD-L1 (nonrandomized).

Note: Cohorts 1 and 2 were closed upon the addition of Cohort 3.

* After TIL growth is established: Patients assigned to Cohort 3 without contraindications to pembrolizumab, will be assigned to receive pembrolizumab in combination with the standard non-myeloblative (NMA) conditioning regimen, TIL, and high-dose IL-s (Arm 2). Patients in Cohort 3 with relative contraindicatioons to prembrolizumab will be assigned to receive standard NMA, TIL, and high dose IL-2 (Arm 3).
* For those patients receiving pembrolizumab- Pembrolizumab will be administered immediately prior to TIL administration and continue for an additional three cycles following the cell infusion.
* Up to 53 patients may be enrolled over 3-4 years.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma with at least one lesion that is resectable for TIL generation.
2. Confirmation of diagnosis of metastatic melanoma by the Laboratory of Pathology of NCI.
3. Patients must have received at least one prior therapy for metastatic melanoma.
4. Patients with 3 or fewer brain metastases that are less than 1 cm in diameter and asymptomatic are eligible. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible.
5. Greater than or equal to 18 years of age and less than or equal to 72 years of age.
6. All participants must sign a written informed consent.
7. All participants must be willing to sign a durable power of attorney
8. Clinical performance status of ECOG 0 or 1.
9. Patients of both sexes must be willing to practice birth control from the time of enrollment on this study and for up to four months after treatment.
10. Serology:

    * Seronegative for HIV antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus are less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
11. Individuals of child-bearing potential must be willing to undergo a pregnancy test prior to the start of treatment because of the potentially dangerous effects of the treatment on the fetus.
12. Individuals of child-bearing potential (IOCBP) must agree to use highly effective contraception (hormonal, intrauterine device [IUD, abstinence, surgical sterilization starting at the time of study entry, for the duration of study therapy, and 12 months after the last dose of combined chemotherapy

    Individuals that can father children must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and for 4 months after the last dose of combined chemotherapy. We also will recommend individuals that can father children ask their partners to be on highly effective birth control (hormonal, intrauterine device (IUD), surgical sterilization).

    NOTE: IOCBP is defined as any female who has experienced menarche and who has not undergone successful surgical sterilization or who is not postmenopausal.

    NOTE: Certain malignancies may secrete hormones that produce false positive pregnancy tests. Serial blood testing (e.g. HCG measurements) and/ or ultrasound may be performed for clarification.

    IOCBP must not donate, or retrieve for their own use, ova from the time of study treatment initiation and throughout the study treatment period, and for at least 12 months after the final study drug(s) administration. Individuals that can father children must not freeze or donate sperm for at least 12 months after the final study drug(s) administration.
13. Nursing participants must be willing to discontinue nursing from study treatment initiation through 4 months after the last dose of the study drug(s).
14. Hematology

    * Absolute neutrophil count greater than 1000/mm3 without the support of filgrastim
    * WBC greater than or equal to 2500/mm3
    * Platelet count greater than or equal to 800,000/mm3
    * Hemoglobin > 8.0 g/dl
15. Chemistry:

    * Serum ALT/AST less than or equal to 2.5 times the upper limit of normal
    * Serum Creatinine less than or equal to 1.6 mg/dl
    * Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert s Syndrome who musthave a total bilirubin less than 3.0 mg/dl.
16. Patients must have completed any prior systemic therapy at the time of enrollment.
17. Patients must demonstrate progressive disease at the time of treatment. (Note: Patients who have received tyrosine kinase inhibitors (e.g. vemurafinib) may be treated if they present with stable disease at the time of treatment).
18. Patients must be co-enrolled in protocol 03-C-0277.

EXCLUSION CRITERIA:

1. Individuals of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
3. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
4. Active systemic infections requiring anti-infective treatment, coagulation disorders or any other active major medical illnesses.
5. History of major organ autoimmune disease
6. Concurrent systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. Grade 3 or 4 Major organ Immune-related Adverse Events (IRAEs) clinically attributed to anti PD-1/PD-L1 monotherapy. Previously screened participants that experience these IRAEs after resection for creation of TIL are excluded from Arms 2, but may be eligible for assignment to Arm3. NOTE: For the purposes of this protocol, thyroid is not considered a major organ.
9. History of coronary revascularization or ischemic symptoms.
10. For select patients with a clinical history prompting cardiac evaluation: last LVEF of less than or equal to 45%
11. For select patients with a clinical history promptin pulmonary evaluation: known FEV1 less than or equal to 50%.
12. Patients who are receiving any other investigational agents.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-12-04 (Actual); Primary Completion 2028-06-16 (Estimated); Study Completion 2029-06-16 (Estimated)

PRIMARY OUTCOMES:
Response rate | 6 and 12 weeks after cell infusion, then every 3 months x3, then every 6 months x 2 years
  Percentage of patients who have a clinical response to treatment (objective tumor regression)

SECONDARY OUTCOMES:
Frequency and severity of treatment-related adverse events | 30 days after end of treatment
  Aggregate of all adverse events, as well as their frequency and severity
Overall survival | Time of death
  Time from start of treatment to death from any cause
Objective response rate (ORR), progression free survival (PFS) and safety (Cohort 3, Arm 3) | 6 and 12 weeks after cell infusion, then every 3 months x 3, then every 6 months x 2 years
  Percentage of patients who have a complete response and/or partial response to treatment
Overall survival (Cohort 3, Arm 3) | Time of death
  Time from start of treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Goff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Rosenberg SA, Yang JC, Sherry RM, Kammula US, Hughes MS, Phan GQ, Citrin DE, Restifo NP, Robbins PF, Wunderlich JR, Morton KE, Laurencot CM, Steinberg SM, White DE, Dudley ME. Durable complete responses in heavily pretreated patients with metastatic melanoma using T-cell transfer immunotherapy. Clin Cancer Res. 2011 Jul 1;17(13):4550-7. doi: 10.1158/1078-0432.CCR-11-0116. Epub 2011 Apr 15. PMID 21498393
- [Background] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Background] Besser MJ, Shapira-Frommer R, Itzhaki O, Treves AJ, Zippel DB, Levy D, Kubi A, Shoshani N, Zikich D, Ohayon Y, Ohayon D, Shalmon B, Markel G, Yerushalmi R, Apter S, Ben-Nun A, Ben-Ami E, Shimoni A, Nagler A, Schachter J. Adoptive transfer of tumor-infiltrating lymphocytes in patients with metastatic melanoma: intent-to-treat analysis and efficacy after failure to prior immunotherapies. Clin Cancer Res. 2013 Sep 1;19(17):4792-800. doi: 10.1158/1078-0432.CCR-13-0380. Epub 2013 May 20. PMID 23690483
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-C-0027.html